CLINICAL TRIAL: NCT05925140
Title: Comparative LUSZ Therapeutic Study of Antiviral, Antiretroviral, and Immunosuppressive Treatments in Hospitalized COVID-19 Patients With High-Risk Factors, Biomarkers, and Disease Progression.
Brief Title: LUSZ Treatment Efficacy in Hospitalized COVID-19 Patients
Acronym: LUSZ_AVIST
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lebanese University (Other)
Collaborators: Hospital Saydet Zgharta University Medical Center (Unknown)
Responsible Party: Principal Investigator, Nehman Makdissy, Principal Investigator, Professor, Lebanese University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVID LUSZ Therapeutic
Record Dates: First submitted 2023-06-28; First posted 2023-06-29 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: COVID-19; Hospitalized COVID-19 Patients
Keywords: Covid-19; SARS-CoV-2; Comorbidities; Score; Inflammation; LUSZ; WHO ordinal severity scale; IL6; Antiviral; Antiretroviral; Immunosuppressive; Therapeutic treatments; Hospitalized COVID-19 patients; High-risk factors; Biomarkers; Disease Progression; Efficacy; Effectiveness; Randomized controlled trial; Treatment outcomes; Survival rates; Mortality; Safety
MeSH Terms: conditions — COVID-19; Inflammation; Disease Progression | interventions — Lopinavir; lopinavir-ritonavir drug combination; remdesivir; tocilizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- LUSZ Control group: Corticosteroid Therapy-enhanced Standard Care (CTSC) alone. (Active Comparator): The control group receives the standard care treatment with corticosteroid therapy.
  Interventions: Other: Corticosteroid Therapy-enhanced Standard Care (CTSC)
- LUSZ Antivirals Group: CTSC + Remdesivir or Lopinavir/Ritonavir. (Experimental): The Antivirals group receives the standard care treatment with corticosteroid therapy in combination with antiviral (Remdesivir) or antiretroviral (Lopinavir/Ritonavir) medications.
  Interventions: Drug: Lopinavir / Ritonavir; Drug: Remdesivir (RDV); Other: Corticosteroid Therapy-enhanced Standard Care (CTSC)
- LUSZ Immunosuppressive Group: CTSC + IL-6 receptor antagonist (Tocilizumab). (Experimental): The Immunosuppressive group receives the standard care treatment with corticosteroid therapy in combination with Tocilizumab, an IL-6 receptor antagonist.
  Interventions: Drug: Tocilizumab; Other: Corticosteroid Therapy-enhanced Standard Care (CTSC)

INTERVENTIONS:
Drug: Lopinavir / Ritonavir — Kaletra is a medication that is produced by AbbVie, a pharmaceutical company based in the United States. It is FDA approved for the treatment of HIV-1 infection in adults and pediatric patients. Kaletra contains two active ingredients, lopinavir, and ritonavir, which work together to inhibit the replication of the HIV virus.
  Administration dose and duration of treatment: Patients will receive a loading dose (800/200, daily) of lopinavir 400 mg plus ritonavir 100 mg orally every 12 h for 10 days or until discharge, if sooner.
  Other Names: Kaletra
  Arms: LUSZ Antivirals Group: CTSC + Remdesivir or Lopinavir/Ritonavir.
Drug: Remdesivir (RDV) — Remdesivir is provided by the United States as an FDA-approved drug, an antiviral medication developed by Gilead Sciences, and has been authorized for emergency use and approved for the treatment of COVID-19 in certain countries, including the United States.
  Administration dose and duration of treatment: intravenously as a 200-mg loading dose on day 1, followed by a 100-mg once daily on days 2-10 or until hospital discharge or death. Duration is generally 5 days or until hospital discharge, whichever is first, but may extend to up to 10 days based on clinical response: For inpatients not requiring IMV and/or ECMO: 5 days; if clinical improvement is not demonstrated, treatment may be extended up to 10 days total. For inpatients requiring IMV and/or ECMO: 10 days.
  Other Names: Veklury
  Arms: LUSZ Antivirals Group: CTSC + Remdesivir or Lopinavir/Ritonavir.
Drug: Tocilizumab — Actemra is an FDA-approved brand name for Tocilizumab, a monoclonal antibody that targets the interleukin-6 (IL-6) receptor, an immunosuppressive drug produced by Roche. It belongs to a class of medications known as IL-6 receptor antagonists and is designed to suppress the activity of the immune system. By blocking IL-6 receptor signaling, Actemra helps reduce inflammation and is used in the treatment of various autoimmune conditions and cytokine release syndrome.
  Administration dose and duration of treatment: TCZ was administered 8 mg/kg intravenously (800 mg per infusion) as a single 60-minute intravenous infusion for 4 Weeks initially. The second infusion (400 mg) after 24 h may be administered based on clinical response in case of respiratory worsening, or 8 mg/kg at T0 followed by 8 mg/kg after 12 h.
  Other Names: Actemra
  Arms: LUSZ Immunosuppressive Group: CTSC + IL-6 receptor antagonist (Tocilizumab).
Other: Corticosteroid Therapy-enhanced Standard Care (CTSC) — (1) Methylprednisone (120mg/24h/IV) followed by 80mg/day (7days), and if necessary, continued with 40mg/day; or a pulse therapy (patient in critical state (360mg/day/IV) for 3 serial days, followed by 80mg/day (7days), and if necessary, continued with a dose of 40mg/day. (2) Standard Care: Normal Saline 0.9% (500cc/24h); vitamins [D (Oravil, 100.000IU/2ml PO STAT), C (10g/250cc in normal saline, 60drops/min/day), B (BECOZYME, 6 ampoules IV STAT)]; Omeprazole (RISEK, 40 mg/day IV); Paracetamol (PREFALGAN, 1g IV each 8h 3 times per day), Ketoprofen (PROFENID, 100mg/12h); Ceftriaxone (ROCEPHIN, 2g/day for 3 consecutive days), Doxycycline (VIBRAMYCIN, 100mg/12h PO for 8 days), Ivermectin (12mg/day for a period of 5 days); TOPLEXIL (Syrup, 10cc/each 8h) or SINECOD (Syrup, 15cc/each 8h); ATORVASTATIN (20mg/day); LOVENOX (40mg/12h if <80kg, or 60mg/12h if >80kg). Tranquillizers: NORMOCALM (400mg/night), XANAX (10mg/day), SEROQUEL (25mg/night), DEPIA (2mg/day), to be administered orally
  Other Names: CTSC

SUMMARY:
This study aims first to assess the efficacy, safety, and effectiveness of the LUSZ COVID-19 therapy consisting of a comparative study of three different treatment approaches: antiviral, antiretroviral, and immunosuppressive IL-6 receptor antagonist, and second to identify high-risk factors and biomarkers associated with fatal outcomes in hospitalized COVID-19 patients. The study seeks to validate a novel predictive scoring model for disease progression and evaluate the impact of these treatments on mortality, admission to the intensive care unit (ICU), and time to recovery.

DETAILED DESCRIPTION:
The ongoing COVID-19 pandemic has posed significant challenges worldwide, necessitating the evaluation of various treatment options to mitigate disease severity and improve patient outcomes. This study aims to conduct a comparative therapeutic analysis of antiviral, antiretroviral, and immunosuppressive treatments in hospitalized COVID-19 patients, named here the COVID-19 LUSZ Therapeutic Stduy. By assessing the efficacy and effectiveness of these treatment modalities, as well as considering high-risk factors, biomarkers, and disease progression, we seek to provide valuable insights into their relative benefits and inform evidence-based therapeutic strategies.

Hypothesis:

Our hypothesis is that certain antiviral, antiretroviral, and immunosuppressive treatments can effectively mitigate disease progression and improve clinical outcomes in hospitalized COVID-19 patients with different degrees of illness severity as classified by the WHO Ordinary Severity Scale (WOSS) adjusted to LUSZ scoring. We postulate that the choice of treatment may depend on the presence of high-risk factors and the underlying immune response, as reflected by biomarker profiles.

Study Design:

This study will adopt a prospective comparative design, analyzing medical records of hospitalized COVID-19 patients from multiple healthcare facilities and evaluating the disease progression. The inclusion criteria will encompass patients diagnosed with COVID-19 and receiving either antiviral, antiretroviral, or immunosuppressive treatments. Patients with comorbidities, varying levels of disease severity, and different treatment durations will be included to reflect real-world clinical scenarios.

Data Collection:

Key variables of interest will include patient demographics, medical history, disease severity at admission, laboratory results, radiology results, treatment regimen, treatment duration, and clinical outcomes. High-risk factors such as advanced age, immunocompromised status, and comorbidities will be specifically analyzed. The pulmonary inflammatory lesion, biomarkers, including inflammatory markers, cytokines, and viral load, will be assessed at various time points to evaluate treatment response and disease progression.

Analysis:

Descriptive statistics will be employed to summarize patient characteristics, treatment modalities, and clinical outcomes. Comparative analysis will be performed to assess the efficacy and effectiveness of antiviral, antiretroviral, and immunosuppressive treatments. Statistical methods, such as chi-square tests, t-tests, Kaplan-Meier survival analysis, and regression analysis, will be utilized to examine associations between treatment regimens and clinical outcomes. Subgroup analyses will be conducted to evaluate treatment response based on high-risk factors and biomarker profiles, applying the LUSZ score.

Targets and Significance:

The primary targets of this study are to compare the therapeutic effects of antiviral, antiretroviral, and immunosuppressive treatments in hospitalized COVID-19 patients and identify potential predictors of treatment response. By elucidating the relative benefits and limitations of these treatment modalities, we aim to contribute to evidence-based clinical decision-making, enhance patient care, and optimize resource allocation. Additionally, this study will provide valuable insights into the interplay between high-risk factors, biomarkers, and disease progression, which can aid in the development of personalized treatment approaches for COVID-19 patients.

In conclusion, this comparative LUSZ therapeutic study in hospitalized COVID-19 patients will provide valuable evidence regarding the efficacy and effectiveness of the LUSZ COVID-19 therapy. By considering high-risk factors, biomarkers, and disease progression, we aim to shed light on the optimal treatment strategies for different patient populations. The findings of this study have the potential to inform clinical practice, improve patient outcomes, and contribute to the ongoing efforts to combat the COVID-19 pandemic.

ELIGIBILITY:
Eligibility Criteria for Hospitalized Patients:

Inclusion criteria:

* Age ≥ 18 years.
* Gender-neutral
* Fulfills WHO case definition, including a positive PCR for COVID-19 from any specimen (e.g., nasopharyngeal, throat, saliva, urine, stool, and other bodily fluid).
* Not received any therapy (radiotherapy, chemotherapy, corticotherapy, hormonotherapy, immunotherapy, anti-inflammatory, antibiotics, antiparasitic, antiviral, antibacterial, convalescent plasma, monoclonal antibodies, or other treatments such as hydroxychloroquine and azithromycin) before admission and samples' collection.
* Spo2 < 90%.
* Moderate to severe COVID-19 cases as defined by WHO ordinal severity scale and clinical and radiological findings.
* The time frame of symptom onset within the past 7 days.
* Participants provide informed consent.
* The study has received ethical approval from the institutional review board: All clinical investigations on human samples will be conducted according to the principles expressed in the Declaration of Helsinki, as revised in 2008 (http://www.wma.net/e/policy/b3.htm). All donors should provide written informed consent, and samples have to be collected in accordance with ethical codes. The study protocol was approved by the institutional review committee of the SZUMC (MA-LE-E-60/2022).

Exclusion criteria:

* Non-SARS-CoV-2.
* Active indication and use of one of the investigational products (e.g., HIV positive if antiretroviral agents were used).
* Allergy or hypersensitivity to one of the investigational products (Lopinavir/Ritonavir, Remdesivir, Tocilizumab) or other contraindication.
* Progression to death is imminent and inevitable within the next 24 hours, irrespective of the provision of treatments.
* Received any therapy (radiotherapy, chemotherapy, corticotherapy, hormonotherapy, immunotherapy, anti-inflammatory, antibiotics, antiparasitic, antiviral, antibacterial, convalescent plasma, monoclonal antibodies, or other treatments such as hydroxychloroquine and azithromycin) before admission and samples' collection.
* Weight loss during the last 2 years.
* Abdominal surgeries.
* Pregnancy.
* SpO2 ≥ 90%.
* Vaccinated individuals were excluded.
* Severe renal impairment (eGFR < 30 mL/min).
* Liver dysfunction (Child-Pugh score ≥ 10).

All included patients should be diagnosed by polymerase chain reaction (PCR) test to be taken from a nasopharyngeal sample, throat sputum, saliva, urine, stool, or bodily fluid. Analyses are to be conducted upon admission as well as 8-10 days after admission. All patients will be followed by the principal investigator of the study. The collection of data from each patient in terms of laboratory data, treatments, and outcomes will be verified by the principal investigator through the review of clinical records. Selected patients will be divided into groups according to the WHO ordinal clinical severity scale.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2020-03-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mortality rate | 28-day mortality rate
  The number of deaths recorded in each arm over a specified period
Clinical improvement rate | 28-day mortality rate
  The proportion of patients showing improvement in clinical symptoms and overall health status in each arm

SECONDARY OUTCOMES:
Time to clinical recovery | 28-day period
  The duration taken for patients to achieve clinical recovery, such as resolution of fever, improvement in respiratory symptoms, and normalization of laboratory markers within 28-day period.
Length of hospital stay | 28-day period
  The number of days patients spend in the hospital from admission to discharge or until a predefined endpoint within a 28-day period.
Disease progression rate | 28-day period
  The rate at which patients experience disease progression, such as the development of severe respiratory distress or organ failure, within a 28-day period.
Adverse events | 28-day period
  The occurrence of any adverse events or side effects related to the treatments in each arm, including drug-related complications or complications associated with immunosuppression, within a 28-day period.
Viral clearance rate | 28-day period
  The rate at which patients in each treatment arm achieve clearance of the SARS-CoV-2 virus from respiratory samples, indicating a reduction in viral replication, within a 28-day period.
Biomarker changes | 28-day period
  Evaluation of changes in specific biomarkers associated with disease severity, inflammation, immune response, or organ dysfunction in each treatment arm within a 28-day period.
Questionnaire about the quality of life | 28-day period
  Assessment of patients' quality of life measures, including physical functioning, psychological well-being, and social aspects, using standardized questionnaires within a 28-day period.
Healthcare resource utilization | 28-day period
  Examination of the utilization of healthcare resources, such as the need for intensive care, mechanical ventilation, or other supportive interventions, in each treatment arm within a 28-day period.

CONTACTS AND LOCATIONS:
Overall Officials: Nehman Makdissy, Professor, Study Chair — Lebanese University
Locations (2):
- Lebanon (2):
  - SZUMC, Zghartā, Mohafazat Liban-Nord
  - Lebanese University, Tripoli

IPD SHARING:
Plan to Share IPD: No